CLINICAL TRIAL: NCT01289457
Title: Phase I/II Randomized Study of Clofarabine, Idarubicin, and Cytarabine (CIA) Versus Fludarabine, Idarubicin, and Cytarabine (FLAI) in Acute Myelogenous Leukemia and High-Risk Myelodysplastic Syndrome
Brief Title: Clofarabine, Idarubicin, and Cytarabine (CIA) Versus Fludarabine, Idarubicin, and Cytarabine (FLAI) in Acute Myelogenous Leukemia (AML) and High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0788; NCI-2011-00251 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: Acute Myelogenous Leukemia; AML; High-Risk Myelodysplastic Syndrome; MDS; Relapsed; Refractory; Clofarabine; Clofarex; Clolar; Idarubicin; Idamycin; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Recurrence | interventions — Clofarabine; Idarubicin; Cytarabine; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Clofarabine + Idarubicin + Cytarabine (Experimental): Phase I: Clofarabine Starting dose 15 mg/m2 by vein for 5 days (days 1-5) + Idarubicin 10 mg/m2 by vein on day 1-3 + Cytarabine 1 g/m2 by vein on day 1-5.
  Interventions: Drug: Clofarabine; Drug: Idarubicin; Drug: Cytarabine; Drug: Fludarabine
- Group 1 CIA (Experimental): Phase II, Group 1 CIA (Clofarabine + Idarubicin + Cytarabine): Clofarabine Maximum Tolerated Dose (MTD) based on Phase I by vein on days 1-5; Idarubicin 10 mg/m2 by vein on days 1-3; Cytarabine 1 g/m2 by vein on days 1-5.
  Interventions: Drug: Clofarabine; Drug: Idarubicin; Drug: Cytarabine
- Group 2 FLAI (Experimental): Phase II, Group 2 FLAI (Fludarabine + Idarubicin + Cytarabine): Fludarabine 30 mg/m2 by vein on days 1-5; Idarubicin 10 mg/m2 by vein on days 1-3; Cytarabine 1 g/m2 by vein on days 1-5.
  Interventions: Drug: Idarubicin; Drug: Cytarabine; Drug: Fludarabine

INTERVENTIONS:
Drug: Clofarabine — Phase I: 15 mg/m2 by vein (IV) daily for 5 days of a 28 day cycle.
  Phase II: Clofarabine (dose selected based on Phase I portion) by vein over approximately 1 hour daily for 5 days (days 1-5) for a 28 day cycle.
  Other Names: Clofarex; Clolar
  Arms: Clofarabine + Idarubicin + Cytarabine; Group 1 CIA
Drug: Idarubicin — 10 mg/m2 by vein over approximately 30 minutes daily for 3 days (days 1-3) of a 28 day cycle.
  Other Names: Idamycin
Drug: Cytarabine — 1 g/m2 by vein over approximately 2 hours daily for 5 days (days 1-5) for a 28 day cycle.
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
Drug: Fludarabine — 30 mg/m2 by vein over approximately 30 minutes daily for 5 days (days 1-5).
  Other Names: Fludara
  Arms: Clofarabine + Idarubicin + Cytarabine; Group 2 FLAI

SUMMARY:
The goal of this clinical research study is to learn if the combination of clofarabine, idarubicin, and cytarabine, or the combination of fludarabine, idarubicin, and cytarabine can help control Acute myeloid leukemia (AML) and Myelodysplastic syndromes (MDS). The safety of these study drug combinations will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Clofarabine is designed to interfere with the growth and development of cancer cells.

Idarubicin is designed to cause breaks in both strands of DNA (the genetic material of cells). This may cause the cancer cells to die.

Cytarabine and Fludarabine are designed to insert themselves into the DNA of cancer cells and stop the DNA from repairing itself.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 4 groups of 6 participants will be enrolled in the Phase I portion of the study. Up to 280 participants will be enrolled in Phase II.

Phase I:

If you are enrolled in the Phase I portion, the dose of clofarabine you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of clofarabine. Each new group will receive a higher dose of clofarabine than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of clofarabine is found.

All participants will receive the same dose level of idarubicin and cytarabine.

Phase II:

If you are enrolled in the Phase II portion, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups:

* If you are in Group 1, you will receive clofarabine, idarubicin, and cytarabine. You will receive clofarabine at the highest dose that was tolerated in the Phase I portion.
* If you are in Group 2, you will receive fludarabine, idarubicin, and cytarabine.

Study Drug Administration:

Study drug(s) will be given in what are called "cycles." Each cycle is 28 days.

Phase I:

On Days 1-5:

* You will receive clofarabine by vein over about 1 hour.
* You will receive cytarabine by vein over about 2 hours.
* On Days 1-3 only, you will receive idarubicin by vein over about 30 minutes.

Phase II (Induction):

The first cycle of study drugs is called Induction. If the doctor thinks it is needed, you will have up to 2 Induction cycles.

If you are in Group 1:

On Days 1-5 of each cycle:

* You will receive clofarabine by vein over about 1 hour.
* You will receive cytarabine by vein over about 2 hours.
* On Days 1-3 only, you will receive idarubicin by vein over about 30 minutes.

If you are in Group 2:

On Days 1-5 of each cycle:

* You will receive fludarabine by vein over about 30 minutes.
* You will receive cytarabine by vein over about 2 hours.
* On Days 1-3 only, you will receive idarubicin by vein over about 30 minutes.

If the doctor thinks it is needed, you may receive less than 5 days of treatment in the induction cycle.

If the doctor thinks it is needed, your dose level will be reduced after Induction.

Phase II (Consolidation):

If the disease responds to the study drugs, you may receive up to 6 more cycles of study drugs. This is called Consolidation.

If you are in Group 1:

On Days 1-3 of each cycle :

* You will receive clofarabine by vein over about 1 hour.
* You will receive cytarabine by vein over about 2 hours.
* After 1 to 2 hours of receiving cytarabine on Days 1-2 only, you will receive idarubicin by vein over about 30 minutes.

If you are in Group 2:

On Days 1-3 of each cycle:

* You will receive fludarabine by vein over about 30 minutes
* You will receive cytarabine by vein over about 2 hours.
* After 1 to 2 hours of receiving cytarabine on Days 1-2 only, you will receive idarubicin by vein over about 30 minutes

If the cancer does not completely respond after Cycle 1, you may repeat induction (Cycle 1). If the cancer completely responds, you will begin the consolidation cycles.

If the doctor thinks it is needed, you may receive less than 3 days of treatment in the consolidation cycles.

Study Visits:

You will have a physical exam, including measurement of your vital signs before the start of each cycle. Blood (about 2 teaspoons) will be drawn for routine tests every 3-7 days.

On Day 28 of every 2-3 cycles (+/- 7 days), if the doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest or up to 8 total cycles. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the long-term follow-up.

Long-Term Follow-up:

Every 3 months for 1 year after you are off study, you will be called and asked how you are feeling, about any side effects you may be having, and about any other drugs you may be taking. These calls should last about 5 minutes each.

This is an investigational study. Cytarabine and Idarubicin are FDA approved and commercially available for the treatment of AML. Fludarabine is FDA approved and commercially available for the treatment of chronic lymphocytic leukemia (CLL). Clofarabine is FDA approved and commercially available for the treatment of acute lymphoblastic leukemia (ALL). The combination of these study drugs is investigational.

Up to 292 patients will take part in Phase I and Phase II of this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an Institutional Review Board (IRB)-approved informed consent document.
2. Age 18 to 60. Patients above the age of 60 only with principal investigator (PI) approval
3. Diagnosis of newly diagnosed AML [other than acute promyelocytic leukemia (APL)] or high-risk (intermediate-2 or high by International Prostate Symptom Score (IPSS) or > 10% blasts, including CMML) MDS. Prior therapy with hydrea and the use of a single or a two day dose of cytarabine (up to 3 g/m2) for emergency use up to 24 hours prior to start of study therapy is allowed. Prior therapy for MDS or other AHD is not allowed.
4. Eastern Cooperative Oncology Group (ECOG) performance status of </= 3 at study entry.
5. Organ function as defined below (unless due to leukemia): Serum creatinine </= 3 mg/dL Total bilirubin </= 2.5 mg/dL , Alanine aminotransferase (ALT) (SGPT) </= 3 * upper limit of normal (ULN) or </= 5 * ULN if related to disease.
6. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days and must agree to practice acceptable contraceptive methods. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.
7. Cardiac ejection fraction >/= 40% (by either cardiac echo or multiple gated acquisition scan (MUGA) scan). Documentation of recent (</= 6 months from screening) outside reports is acceptable.

Exclusion Criteria:

1. Breast feeding females
2. Patients with uncontrolled active infections (viral, bacterial, and fungal are not eligible).
3. Patients with active secondary malignancy will not be eligible.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 282 (Actual)
Dates: Start 2011-02-02 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Morita K, Kantarjian HM, Wang F, Yan Y, Bueso-Ramos C, Sasaki K, Issa GC, Wang S, Jorgensen J, Song X, Zhang J, Tippen S, Thornton R, Coyle M, Little L, Gumbs C, Pemmaraju N, Daver N, DiNardo CD, Konopleva M, Andreeff M, Ravandi F, Cortes JE, Kadia T, Jabbour E, Garcia-Manero G, Patel KP, Futreal PA, Takahashi K. Clearance of Somatic Mutations at Remission and the Risk of Relapse in Acute Myeloid Leukemia. J Clin Oncol. 2018 Jun 20;36(18):1788-1797. doi: 10.1200/JCO.2017.77.6757. Epub 2018 Apr 27. PMID 29702001
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine + Idarubicin + Cytarabine: Phase I: Clofarabine Starting dose 15 mg/m2 by vein for 5 days (days 1-5) + Idarubicin 10 mg/m2 by vein on day 1-3 + Cytarabine 1 g/m2 by vein on day 1-5.
  Clofarabine: Phase I: 15 mg/m2 by vein (IV) daily for 5 days of a 28 day cycle.
  Phase II: Clofarabine (dose selected based on Phase I portion) by vein over approximately 1 hour daily for 5 days (days 1-5) for a 28 day cycle.
  Idarubicin: 10 mg/m2 by vein over approximately 30 minutes daily for 3 days (days 1-3) of a 28 day cycle.
  Cytarabine: 1 g/m2 by vein over approximately 2 hours daily for 5 days (days 1-5) for a 28 day cycle.
- Group 1 CIA: Phase II, Group 1 CIA (Clofarabine + Idarubicin + Cytarabine): Clofarabine MTD based on Phase I by vein on days 1-5; Idarubicin 10 mg/m2 by vein on days 1-3; Cytarabine 1 g/m2 by vein on days 1-5.
  Clofarabine: Phase I: 15 mg/m2 by vein (IV) daily for 5 days of a 28 day cycle.
  Phase II: Clofarabine (dose selected based on Phase I portion) by vein over approximately 1 hour daily for 5 days (days 1-5) for a 28 day cycle.
  Idarubicin: 10 mg/m2 by vein over approximately 30 minutes daily for 3 days (days 1-3) of a 28 day cycle.
  Cytarabine: 1 g/m2 by vein over approximately 2 hours daily for 5 days (days 1-5) for a 28 day cycle.
Period: Overall Study
Arm/Group | Clofarabine + Idarubicin + Cytarabine | Group 1 CIA | Group 2 FLAI
Started | 12 | 157 | 113
Completed | 12 | 157 | 113
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clofarabine + Idarubicin + Cytarabine | Group 1 CIA | Group 2 FLAI | Total
Number analyzed (Participants) | 12 | 157 | 113 | 282
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 153 | 108 | 272
  >=65 years | 1 | 4 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 52 [27 to 68] | 53 [20 to 68] | 51 [18 to 69] | 53 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 74 | 55 | 135
  Male | 6 | 83 | 58 | 147
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 6 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 20 | 11 | 34
  White | 8 | 122 | 85 | 215
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 12 | 157 | 113 | 282

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Clofarabine, Idarubicin, and Cytarabine
Description: MTD is highest dose level in which <2 patients of 6 develop first cycle dose limiting toxicities (DLT). Toxicity defined as any treatment-related grade 3 or greater non-hematological toxicities.
Time Frame: 28 days
Population: Maximum Tolerated Dose (MTD) is only reported for the Phase I portion of the study. MTD was not done on the Phase II portion of the study and therefore, PhII Groups 1 and 2 do not have results for MTD.
Measure: Number; unit: mg/m^2
Arm/Group | Clofarabine + Idarubicin + Cytarabine | Group 1 CIA | Group 2 FLAI
Number analyzed (Participants) | 12 | 0 | 0
mg/m^2 | 15 |  |

2. Secondary Outcome: Response Rates of Clofarabine, Idarubicin, and Cytarabine (CIA) Versus Fludarabine, Idarubicin, and Cytarabine (FLAI)
Description: NCI & Myelodysplastic syndromes (MDS) International Working Group (IWG) Definitions: Complete Response (CR): Neutrophil count ≥1.0 ×10^9/L, Platelet count ≥100 ×10^9/L, Bone marrow aspirate </=5% blasts, No extramedullary leukemia; CRi: Response as in CR but platelets <100 ×10^9/L; Partial response (PR): Neutrophil count ≥ 1.0 ×10^9/L, Platelet count ≥100 ×10^9/L, ≥ 50% reduction in bone marrow blasts over baseline; Clinical benefit: In addition to IWG criteria, in AML, a decrease in bone marrow blasts to <5% is also considered clinical benefit; Stable Disease: In addition to IWG criteria and in absence any of above response criteria, stable disease considered if the bone marrow blast percent does not increase compared to pretreatment level; Relapse: Increase of bone marrow blasts to >10% after initial response. Response assessed Day 28 of every 2-3 cycles during treatment.
Time Frame: 12 months
Population: The outcome measure for for the Phase I portion of this study was to determine MTD only. Data Was not collected for Response Rate for the Phase I arm of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine + Idarubicin + Cytarabine | Group 1 CIA | Group 2 FLAI
Number analyzed (Participants) | 0 | 157 | 113
Participants |  | 107 | 76

3. Secondary Outcome: Event-Free Survival (EFS) at 2 Years
Description: Comparison of the event-free survival (EFS) between treatment CIA and FLAI, where an event is defined to be resistance to treatment, relapse (after response) or death, whichever occurred first.
Time Frame: Up to 2 years or until relapse/death
Population: The outcome measure for for the Phase I portion of this study was to determine MTD only. Data Was not collected for EFS for the Phase I arm of this study.
Measure: Median (Full Range); unit: Months
Arm/Group | Clofarabine + Idarubicin + Cytarabine | Group 1 CIA | Group 2 FLAI
Number analyzed (Participants) | 0 | 157 | 113
Months |  | 7.1 [1 to 69] | 8.4 [1 to 69]

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: up to 2 years
Population: The outcome measure for the Phase I portion of this study was to determine MTD only. Data Was not collected for Overall Survival for the Phase I arm of this study.
Measure: Median (Full Range); unit: Months
Arm/Group | Clofarabine + Idarubicin + Cytarabine | Group 1 CIA | Group 2 FLAI
Number analyzed (Participants) | 0 | 157 | 113
Months |  | 14.5 [1 to 70] | 15.1 [1 to 70]

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Clofarabine + Idarubicin + Cytarabine | Group 1 CIA | Group 2 FLAI
All-Cause Mortality (participants affected / at risk) | 4/12 | 8/157 | 5/113
Serious Adverse Events (participants affected / at risk) | 10/12 | 126/157 | 89/113
Other Adverse Events (participants affected / at risk) | 12/12 | 150/157 | 109/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Idarubicin + Cytarabine (N=12) | Group 1 CIA (N=157) | Group 2 FLAI (N=113)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Allergic Reaction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Altered Mental Status (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bell's Palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 0 | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 4 (4) | 5 (5) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Disseminated Intravastular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Drain Placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Elevated Alanine Aminotransferase (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (2)
Elevated Amylase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated Amylase/Lipase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Elevated Lipase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 4 (4) | 3 (3)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 6 (7) | 8 (8)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (General disorders) | 7 (9) | 52 (80) | 23 (26)
Kidney Stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Mental Status (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (7) | 5 (7)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenic Fever (Infections and infestations) | 2 (2) | 75 (122) | 57 (88)
Pain (General disorders) | 0 (0) | 12 (15) | 12 (16)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Idarubicin + Cytarabine (N=12) | Group 1 CIA (N=157) | Group 2 FLAI (N=113)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5)
Mental Status (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Hemorrhage CNS (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 2 (2)
CNS Cerebrovascular Ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syndromes Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (10) | 1 (1)
Elevated Creatinine (Metabolism and nutrition disorders) | 0 (0) | 10 (10) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 9 (9) | 5 (5)
Hemorrhage, Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 4 (5) | 7 (9)
Hypotension (Cardiac disorders) | 1 (1) | 8 (9) | 4 (4)
Opportunistic Infection (Infections and infestations) | 0 (0) | 6 (7) | 7 (7)
Elevated Aspartate Aminotransferase (Metabolism and nutrition disorders) | 2 (2) | 17 (17) | 4 (4)
Anorexia (Gastrointestinal disorders) | 0 (0) | 18 (18) | 13 (13)
Vomiting (Gastrointestinal disorders) | 0 (0) | 23 (27) | 9 (11)
Mucositis/Stomatitis (Gastrointestinal disorders) | 0 (0) | 23 (24) | 12 (15)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 29 (29) | 20 (20)
Fatigue (General disorders) | 1 (1) | 29 (30) | 21 (22)
Elevated Alanine Aminotransferase (Metabolism and nutrition disorders) | 2 (2) | 40 (42) | 11 (11)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 7 (7) | 40 (42) | 11 (11)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 43 (47) | 14 (14)
Nausea (Gastrointestinal disorders) | 1 (1) | 42 (45) | 27 (29)
Pain (General disorders) | 0 (0) | 43 (53) | 24 (29)
Neutropenic Fever (Infections and infestations) | 8 (9) | 94 (140) | 48 (80)
Infection (Infections and infestations) | 11 (29) | 70 (136) | 39 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT01289457/Prot_SAP_000.pdf